CLINICAL TRIAL: NCT06065631
Title: Seeing to Learn in Sierra Leone: Impact of Spectacle Correction on Children's Academic Performance and Mental Health Wellbeing
Brief Title: Seeing to Learn in Sierra Leone
Acronym: SLII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: USAID stopped funding the study in March of 2025 because USAID was dismantled and stopped funding all research programs.
Sponsor: University of Minnesota (Other)
Collaborators: Innovations for Poverty Action (Other); Peek Vision (Unknown); Vision Action (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Glewwe Transfer
Record Dates: First submitted 2023-09-21; First posted 2023-10-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Refractive Errors
Keywords: Myopia; Hyperopia; Spectacle correction; Educational outcomes
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia | interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: All eligible children will be randomized by school to receive at the start of the school year either: free ready-made or custom eyeglasses (Intervention), or an eyeglasses prescription and letter to parents, with free eyeglasses at endline (Control). The clusters (schools) will be stratified into groups based on the prevalence of refractive error and on the score on the baseline mathematics and reading exams. The division of the sample into schools in the two cities (Bo and Freetown) will be in the same proportion as the proportion of the number of public schools in those two cities.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be given either glasses or a prescription. Hence, they could not be masked.
  The Care Provider, in our case, screening and examination team will be providing either glasses or prescriptions to the participants. Hence, they could not masked.
  Investigators and Outcome assessor will only analyse the data at the end of the trial and they will not be
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): An eyeglasses prescription and letter to parents, with free eyeglasses at endline.
  Interventions: Other: Prescription slip
- Intervention (Experimental): free ready-made or custom eyeglasses
  Interventions: Device: Eyeglasses

INTERVENTIONS:
Device: Eyeglasses — Children with uncorrected/under-corrected refractive error will be provided with either ready made or custom eyeglasses based on their magnitude and types of refractive errors.
  Other Names: Glasses; Spectacle
  Arms: Intervention
Other: Prescription slip — Children with uncorrected/under-corrected refractive error will be provided with an eyeglasses prescription and letter to parents, but all of them will get eyeglasses at the end of the trial
  Arms: Control

SUMMARY:
The main objective of the Sierra Leone Sees to Learn (SL2) trial is to assess the educational impact of providing free eyeglasses to students aged 9-20 years with uncorrected refractive error in Sierra Leone. The procedures include baseline questionnaires and educational assessments to collect data on students and schools, and then the provision of free eyeglasses to students who have uncorrected (or undercorrected) refractive error (URE). The questionnaires and student assessments will take 1-2 hours. The duration of the study timeframe is one school year. The end-line questionnaires and student assessments will be administered at the end of the school year.

DETAILED DESCRIPTION:
Objective: The main objective of the Sierra Leone Sees to Learn (SL2) trial is to assess the educational impact of providing free eyeglasses to students aged 9-20 years with uncorrected refractive error in Sierra Leone.

Sample frame: Approximately 2400 children with uncorrected (or undercorrected) refractive error (URE) at 300 randomly-selected schools in Freetown and Bo City. A similar number of children from the same schools but without vision problems will also be included, at baseline only, to compare their basic demographic characteristics and daily activities to those of the children with URE. The sample size may vary depending on the percentage of children with URE obtained from screening a total of 40,000 children. All children with URE as specified in the enrolment criteria below will be part of the study.

Design: Cluster-randomized control trial (cluster RCT), with schools as clusters.

Randomization, interventions and balancing: All eligible children will be randomized by school to receive at the start of the school year either: free ready-made or custom eyeglasses (Intervention), or an eyeglasses prescription and letter to parents, with free eyeglasses at end-line (Control). The clusters (schools) will be stratified into groups based on the prevalence of refractive error and on the score on the baseline mathematics and reading exams. The division of the sample into schools in the two cities (Bo and Freetown) will be in the same proportion as the proportion of the number of public schools in those two cities.

Power calculations (reading and math exams): Setting power = 0.8, statistical precision = 0.05, intracluster correlation = 0.2 (from 2019 Sierra Leone grade 8 learning assessment), 80 treated schools, 80 control schools, 15 students/school with uncorrected error, yields the following minimal detectable effect (MDE) sizes as a function of correlation between baseline and end-line tests:

MDE Correlation of baseline and end-line tests 0.101 0.7 0.127 0.6 0.148 0.5

A nested focus-group study will explore children's, parents' and teachers' attitudes towards vision, student learning, and wearing of eyeglasses, in order to design a locally-tailored intervention to promote wearing of eyeglasses.

Regression Framework:

The investigators will estimate the effect of the program using a single difference cross-sectional ordinary least squares regression (OLS), and a difference-in-difference (DID) OLS regression that includes observations at both end-line and baseline. The investigators will report two types of effects: the intent-to-treat (ITT) effects and local average treatment effects (LATE), using treatment assignment as an instrumental variable for participation. Analysis will use the observed baseline characteristics as control variables and account for school-level variation through a fixed effect.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting (with or without glasses) distance visual acuity of 6/12 or worse in the better-seeing eye;
2. Refractive error of at least 0.75 diopters (D) of myopia, 2.00 D of hyperopia or 1.00 D of astigmatism;
3. Visual acuity is correctable to 6/7.5 or better with eyeglasses.

Exclusion Criteria:

1. Other ocular problems preventing visual acuity > 6/12 in both eyes.

Ages: 9 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1821 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Foundational mathematic and literacy skills | Month 1 and 9 months after glasses are provided
  Item Response Theory to estimate a student's ability on a continuous scale and subsequently standardize students' scores on a continuous scale with respect to the control-group distribution at baseline (mean zero, standard deviation of one). Lower scores will indicate lower performance, and higher scores will indicate higher performance. A -1 would indicate a student's performance is 1 standard deviation below the mean of the control-group performance distribution at baseline. A zero would mean the student performed like the mean student in the control group at baseline.
Anxiety | Month 1 and 9 months after glasses are provided
  Measured using Generalized Anxiety Disorder 2-item (GAD-2) questionnaire, the highest score is 8 and the lowest score is 2. Higher scores indicated more severe anxiety disorders.
Prosocial | Month 1 and 9 months after glasses are provided
  Measured using Strengths & Difficulties Questionnaire with the prosocial score ranges from 0 to 10 and higher scores indicate more prosocial behaviour.
Social and emotional problems | Month 1 and 9 months after glasses are provided
  Measured using Strengths & Difficulties Questionnaire with the score ranges from 0 to 40. Higher scores indicate more social and emotional problems.

SECONDARY OUTCOMES:
Teacher-observed wearing of eyeglasses of children | Month 1 to Month 9 after glasses are provided
  Proportion of children observed wear across all children at daily assessments
Self-reported wearing of eyeglasses compliance | Month 9 after glasses are provided
  Proportion of children who reported to be wearing their eyeglasses 1. Not at all 2. Sometimes 3. Most of the time 4. All the time
Enumerator-observed wearing of eyeglasses | At Months 3, 6 and 9 after glasses are provided
  Actual presence of spectacles on the child's face (rather than having glasses at school) at the time of an unannounced examination
Cost-effectiveness 1 | Through study completion, an average of 9 months
  Total eyeglasses distribution cost (excluding study cost) per child receiving, and wearing, eyeglasses at endline
Cost-effectiveness 2 | Through study completion, an average of 9 months
  Total eyeglasses distribution cost (excluding study cost) per 0.1 standard deviation test score gain
School attendance | Daily from Month 1 to Month 9
  Attendance data will be collected from attendance registry at school. This will be expressed in percentage. Lowest attendance being 0%, highest being 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Innovations for Poverty Action (IPA), Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: Yes
Only deidentified data will be shared, on request.
Supporting Information: SAP
Time Frame: Data will be available once they are cleaned and de-identified, kept for at least 10 years after study completion
Access Criteria: Those who wish to access the de-identified data will need to request formally with the research team.

REFERENCES:
- [Result] GBD 2019 Blindness and Vision Impairment Collaborators; Vision Loss Expert Group of the Global Burden of Disease Study. Trends in prevalence of blindness and distance and near vision impairment over 30 years: an analysis for the Global Burden of Disease Study. Lancet Glob Health. 2021 Feb;9(2):e130-e143. doi: 10.1016/S2214-109X(20)30425-3. Epub 2020 Dec 1. PMID 33275950
- [Result] Burton MJ, Ramke J, Marques AP, Bourne RRA, Congdon N, Jones I, Ah Tong BAM, Arunga S, Bachani D, Bascaran C, Bastawrous A, Blanchet K, Braithwaite T, Buchan JC, Cairns J, Cama A, Chagunda M, Chuluunkhuu C, Cooper A, Crofts-Lawrence J, Dean WH, Denniston AK, Ehrlich JR, Emerson PM, Evans JR, Frick KD, Friedman DS, Furtado JM, Gichangi MM, Gichuhi S, Gilbert SS, Gurung R, Habtamu E, Holland P, Jonas JB, Keane PA, Keay L, Khanna RC, Khaw PT, Kuper H, Kyari F, Lansingh VC, Mactaggart I, Mafwiri MM, Mathenge W, McCormick I, Morjaria P, Mowatt L, Muirhead D, Murthy GVS, Mwangi N, Patel DB, Peto T, Qureshi BM, Salomao SR, Sarah V, Shilio BR, Solomon AW, Swenor BK, Taylor HR, Wang N, Webson A, West SK, Wong TY, Wormald R, Yasmin S, Yusufu M, Silva JC, Resnikoff S, Ravilla T, Gilbert CE, Foster A, Faal HB. The Lancet Global Health Commission on Global Eye Health: vision beyond 2020. Lancet Glob Health. 2021 Apr;9(4):e489-e551. doi: 10.1016/S2214-109X(20)30488-5. Epub 2021 Feb 16. No abstract available. PMID 33607016
- [Result] Dandona L, Dandona R. What is the global burden of visual impairment? BMC Med. 2006 Mar 16;4:6. doi: 10.1186/1741-7015-4-6. PMID 16539747
- [Result] Glewwe P, West KL, Lee J. The Impact of Providing Vision Screening and Free Eyeglasses on Academic Outcomes: Evidence from a Randomized Trial in Title I Elementary Schools in Florida. J Policy Anal Manage. 2018;37(2):265-300. doi: 10.1002/pam.22043. PMID 29693366
- [Result] Keil S, Fielder A, Sargent J. Management of children and young people with vision impairment: diagnosis, developmental challenges and outcomes. Arch Dis Child. 2017 Jun;102(6):566-571. doi: 10.1136/archdischild-2016-311775. Epub 2016 Nov 16. PMID 27852581
- [Result] Ma X, Zhou Z, Yi H, Pang X, Shi Y, Chen Q, Meltzer ME, le Cessie S, He M, Rozelle S, Liu Y, Congdon N. Effect of providing free glasses on children's educational outcomes in China: cluster randomized controlled trial. BMJ. 2014 Sep 23;349:g5740. doi: 10.1136/bmj.g5740. PMID 25249453
- [Result] Naidoo KS, Raghunandan A, Mashige KP, Govender P, Holden BA, Pokharel GP, Ellwein LB. Refractive error and visual impairment in African children in South Africa. Invest Ophthalmol Vis Sci. 2003 Sep;44(9):3764-70. doi: 10.1167/iovs.03-0283. PMID 12939289
- [Result] Ma Y, Congdon N, Shi Y, Hogg R, Medina A, Boswell M, Rozelle S, Iyer M. Effect of a Local Vision Care Center on Eyeglasses Use and School Performance in Rural China: A Cluster Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jul 1;136(7):731-737. doi: 10.1001/jamaophthalmol.2018.1329. PMID 29801081
- [Result] Wang X, Yi H, Lu L, Zhang L, Ma X, Jin L, Zhang H, Naidoo KS, Minto H, Zou H, Rozelle S, Congdon N. Population Prevalence of Need for Spectacles and Spectacle Ownership Among Urban Migrant Children in Eastern China. JAMA Ophthalmol. 2015 Dec;133(12):1399-406. doi: 10.1001/jamaophthalmol.2015.3513. PMID 26426113
- [Result] Williams WR, Latif AH, Hannington L, Watkins DR. Hyperopia and educational attainment in a primary school cohort. Arch Dis Child. 2005 Feb;90(2):150-3. doi: 10.1136/adc.2003.046755. PMID 15665167